CLINICAL TRIAL: NCT03994549
Title: A First in Human, Randomized, Double-blind, Placebo-controlled, Single Ascending Dose Trial Assessing Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of a Single Subcutaneous Dose of ZP7570 in Healthy Subjects
Brief Title: A Single Ascending Dose Trial Assessing Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of ZP7570
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Zealand Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ZP7570-18144; 2019-001128-36 (EudraCT Number)
Record Dates: First submitted 2019-05-15; First posted 2019-06-21 (Actual); Last update posted 2020-12-02 (Actual); Status verified 2020-11

CONDITIONS: Healthy
Keywords: Dual GLP-1R/GLP-2 Receptor agonist

STUDY DESIGN:
Intervention Model Description: A randomized, double-blind, placebo-controlled, single ascending dose trial in healthy subjects, randomized to ZP7570 or placebo
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ZP7570 (Active Comparator): Single subcutaneous injection
  Interventions: Drug: Dual GLP-1/GLP-2 Receptor agonists
- Placebo (Placebo Comparator): Single subcutaneous injection
  Interventions: Drug: Dual GLP-1/GLP-2 Receptor agonists

INTERVENTIONS:
Drug: Dual GLP-1/GLP-2 Receptor agonists — Eight ascending doses of ZP7570
  Other Names: ZP7570

SUMMARY:
This is a randomized, double-blind, placebo-controlled, single ascending dose trial in healthy subjects, randomized to ZP7570 or placebo within each cohort.

DETAILED DESCRIPTION:
Sixty-four subjects are planned to be studied in eight cohorts in this first-in human trial. Eight subjects will be allocated to the to eight dose levels. The entire observation period comprise 28 days starting with a 96 hours in-house stay, where discharge is planned for Day 5, followed by five outpatient visits and an End of Trial Visit at Day 28. A blinded evaluation of each cohort will be performed by a Trial Safety Group to determine whether the trial will progress to the next dose level based on the stopping rules specified in protocol.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or female subject aged between 18 and 55 years, both inclusive.
* Body Mass Index (BMI) between 18.5 and 28.0 kg/m^2, both inclusive
* Body weight of at least 60 kg.
* Heart rate after 5 minutes rest in supine position inside the range of 50-90 beats/min at screening

Exclusion Criteria:

* Any history of a disorder which in the investigator's opinion might jeopardize subjects safety, evaluation of results or compliance with the protocol.
* History of gallbladder disease or cholecystectomy.
* History of major depressive disorder or a Patient Health Questionnaire (PHQ-9) > 9 completed at screening, or a history of other severe psychiatric disorders (e.g. schizophrenia or bipolar disorder).
* Any suicidal ideation of type 4 or 5 on the Columbia-Suicide Severity Rating Scale (C-SSRS) within 6 months prior to screening.
* Clinically significant abnormal standard 12-lead ECG after 5 min resting in supine position at screening, including a QTcF > 450 ms (males) or QTcF > 470 ms (females), PR ≥ 220 ms and QRS ≥ 110 ms as evaluated by the investigator.
* History of severe hypersensitivity to medicines or foods or history of severe medicinal/food induced anaphylactic reaction or contraindication to the use of Indocyanine Green (e.g. hypersensitivity to iodine).
* Any clinically significant abnormal hematology, biochemistry, or urinalysis screening tests, as judged by the investigator.
* TSH values outside of normal reference ranges of safety laboratory
* Estimated glomerular filtration rate (eGFR) < 90 ml/min/1.73 m2, as defined by Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI).
* Known or suspected hypersensitivity to IMP(s) or related products.
* Systolic blood pressure < 90 mmHg or >139 mmHg and/or diastolic blood pressure < 50 mmHg or > 89 mmHg (one repeat test will be acceptable in case of suspected white-coat hypertension).
* Symptoms of arterial hypotension
* Women of childbearing potential who are not using a highly effective contraceptive method
* Men with non-pregnant partner(s) of childbearing potential not willing to use male contraception (condom) in addition to a highly effective contraceptive method until 28 days after dosing
* Men with pregnant partner not willing to use male contraception (condom) until 28 days after dosing, in order to avoid exposure of the embryo/fetus to seminal fluid

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 64 (Actual)
Dates: Start 2019-06-14 (Actual); Primary Completion 2020-11-02 (Actual); Study Completion 2020-11-02 (Actual)

PRIMARY OUTCOMES:
Safety - Incidence of adverse events (AEs) | From time zero to 28 days after dosing
  The incidence, type and severity of adverse events (AEs)

SECONDARY OUTCOMES:
Pharmacokinetics - Area under the plasma concentration-time curve trough | From time zero up to day 28
  AUCτ, Area under the plasma concentration-time curve (AUC) from zero up to trough concentration.
Pharmacokinetics - Area under the plasma concentration-time curve infinity | From time zero up to day 28
  AUCinf, Area under the plasma concentration-time curve (AUC) from zero up to last concentration.
Pharmacokinetics - Area under the plasma concentration-time curve last | From time zero up to day 28
  AUClast, Area under the plasma concentration-time curve (AUC) from zero up to last concentration
Pharmacokinetics - Maximum plasma concentration | From time zero to 28 days after dosing
  Measured maximum plasma drug concentration after dosing, Cmax
Pharmacokinetics - Time to maximum plasma concentration (Tmax) | From time zero to 28 days after dosing
  Sampling time until reaching Cmax, Tmax
Pharmacokinetics - Half-life , t½ | From time zero to 28 days after dosing
  Half-life of ZP7570, t½
Pharmacokinetics - Volume of distribution | From time zero to 28 days after dosing
  Apparent volume of distribution of ZP7570, Vz/f
Pharmacokinetics - Mean residence time | From time zero to 28 days after dosing
  Mean residence time, MRT
Pharmacokinetics - Body clearance | From time zero to 28 days after dosing
  Total body clearance, CL/f
Pharmacokinetics - Elimination rate constant | From time zero to 28 days after dosing
  Elimination rate constant, λz
Pharmacodynamics - Plasma glucose levels | Time Frame: 0-240 minutes
  Plasma glucose levels included with the acetaminophen at specific timepoints relative to a Mixed Test Meal
Pharmacodynamics - Insulin concentrations | Time Frame: 0-240 minutes
  Insulin concentrations included with the acetaminophen at specific timepoints relative to a Mixed Test Meal
Pharmacodynamics - Plasma acetaminophen concentration-time curves | Time Frame: 0-240 minutes
  Plasma acetaminophen concentration-time curves following ingestion of acetaminophen
Pharmacodynamics - Maximum acetaminophen concentration | Time Frame: 0-240 minutes
  Change from baseline acetaminophen to maximum acetaminophen
Pharmacodynamics - Time maximum acetaminophen concentration | Time Frame: 0-240 minutes
  Time to maximum change in acetaminophen measure from baseline, Tmax
Safety - Safety lab, haematology | From time zero to 28 days after dosing
  Changes in haematology parameters: Haematocrit, Haemoglobin, Erythrocytes, MCV, MCH, MCHC, platelets, Leucocytes, Neutrophile granulocytes (total count and relative), Lymphocytes (total count and relative), Monocytes (total count and relative), Eosinophile granulocytes (total count and relative), Basophile granulocytes (total count and relative)
Safety - Safety lab, clinical chemistry | From time zero to 28 days after dosing
  Changes in clinical chemistry parameters: Sodium, Potassium, Calcium, Creatinine, Urea, AST, ALT, gamma-GT, Uric acid, Total protein, Albumin, Total bilirubin, Creatine kinase, Alkaline phosphatase, LDH, Total cholesterol, LDL, HDL, Amylase, Triglycerides, Lipase
Safety - Safety lab, urinalysis | From time zero to 28 days after dosing
  Changes in urinalysis: Protein, Glucose Erythrocytes, Leucocytes, pH, ketones
Safety - Vital signs, blood pressure | From time zero to 28 days after dosing
  Changes in vital signs, blood pressure (in mmHG)
Safety - Vital signs, pulse | From time zero to 28 days after dosing
  Changes in pulse (beats per minute)
Safety - Physical examination | From time zero to 28 days after dosing
  Changes in physical examination of body sections (head, chest and heart, abdomen, skin and mucosae, musculoskeletal system, nervous system, lymph node)
Safety - ECG | From time zero to 28 days after dosing
  Occurrence of ECG findings, Changes in ECG parameters (in ms). ECG components: Heart rate, PR, QRS, QT and QTcF.
Safety - Occurrence of Injection site reactions | From time zero to 28 days after dosing
  Occurrence of injection site reactions
Safety - Immunogenicity: Occurrence of anti-drug antibodies | From time zero to 28 days after dosing
  Occurrence of anti-drug antibodies

CONTACTS AND LOCATIONS:
Overall Officials: Ulrike Hövelmann, MD, Principal Investigator — Profil Neuss, Germany
Locations (1):
- Profil Institut für Stoffwechselforschung GmbH, Neuss, North Rhine-Westphalia, Germany

IPD SHARING:
Plan to Share IPD: No